CLINICAL TRIAL: NCT03689439
Title: Is Bone Scintigraphy Necessary in cT1N0M0 GGO Non-Small Cell Lung Cancer?
Brief Title: Is Bone Scintigraphy Necessary in cT1N0M0 GGO Non-Small Cell Lung Cancer? (ECTOP-1006)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Other Study IDs: ECTOP-1006
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Bone Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: bone scintigraphy — bone scintigraphy

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1006. In this prospective one-arm observational study, bone scintigraphy will be performed in T1N0M0 NSCLC patients with GGO lesion and other low risk factors of bone metastasis. The occurrence rate of bone metastasis in these patients will be analyzed to evaluate the necessity of bone scintigraphy in cT1N0M0 NSCLC patients.

DETAILED DESCRIPTION:
Skeletal is a common metastatic site in patients with non-small cell lung cancer. The incidence of bone metastases is about 20-30％ in NSCLC patients. According to the NCCN guidelines, early lung cancer patients should also undergo bone scan or PETCT before surgery to determine the presence of bone metastases. However, all of the above methods use radionuclide reagents as tracers, which pose health hazards to patients and their contacts, including medical personnel. A retrospective study conducted by our center showed that only 0.95% of patients with cT1N0M0 non-small cell lung cancer had preoperative bone metastases. In patients with early stage lung cancer whose lesions are pure ground glass nodules, the probability of developing bone metastases is zero. The low risk factors for bone metastases from this retrospective study included preoperative examination of patients with CEA <5 ng/ul and no bone-related symptoms. In patients with primary NSCLC who underwent CEA <5 ng/ul preoperatively, no bone metastases occurred; in patients with negative bone-related symptoms, the incidence of bone metastases was only 0.18%. In the case of such patients, if the bone scan is performed, not only the potential damage to the patient is increased, but also the waste of medical resources and the burden on the patient from the perspective of health economics.

Therefore, our center is expected to conduct this prospective one-arm observational clinical trial. According to the low-risk factors derived from retrospective studies, bone scintigraphy was performed in patients with GGO lesion and other low risk factors of bone metastasis, and the incidence of bone metastasis was obtained. The necessity of bone scintigraphy in cT1N0M0 NSCLC patients would be evaluated.

This trial is recognizes in our institute as "Eastern Cooperative Thoracic Oncology Project (ECTOP-1006)"

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form and are willing to complete the study according to the plan;
2. Age 18-80 years old;
3. ECOG score ≤ 2 points;
4. CT shows that the main lesion is considered to be ground glass nodular lung cancer;
5. Preoperative examination CEA <5ng/ul
6. There are no bone related symptoms
7. There is no obvious absolute surgical contraindication for preoperative examination.

Exclusion Criteria:

1. History of bone related diseases.
2. History of other kinds of cancer

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cT1N0M0 NSCLC Patients
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The Occurrence Rate of Bone metastasis in cT1N0M0 NSCLC patients | 1 month
  The Number of cT1N0M0 NSCLC patients that had bone metastasis in this cohort

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, Ph.D, Principal Investigator — Shanghai Cancer Center
Locations (5):
- China (5):
  - Anhui Chest Hospital, Hefei, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiang Du People's Hospital, Yangzhou, Jiangsu
  - Fudan University Cancer Center, Shanghai, Shanghai Municipality
  - Jilin Cancer Hospital, Changchun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li H, Ye T, Li N, Xia G, Li B, Zhang Y, Hu H, Sun Y, Zhang Y, Xiang J, Ma D, Weng Y, Liu S, Jia C, Qian B, Gu Y, Li Y, Song S, Chen H. Is 99m Tc bone scintigraphy necessary in the preoperative workup for patients with cT1N0 subsolid lung cancer? A prospective multicenter cohort study. Thorac Cancer. 2021 Feb;12(4):415-419. doi: 10.1111/1759-7714.13752. Epub 2020 Nov 19. PMID 33210466